CLINICAL TRIAL: NCT04230707
Title: The Role of Endogenous Melatonin Levels on Preoperative and Postoperative Anxiety in Living Liver Donors
Brief Title: Endogenous Melatonin Levels on Anxiety in Living Liver Donors
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Inonu University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Mehmet Ali Erdoğan, Prof.Dr. Mehmet Ali Erdogan, Inonu University
Other Study IDs: MAE6; 217S871 (Registry Identifier: TÜBİTAK)
Record Dates: First submitted 2019-10-14; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Liver Transplantation; Anxiety; Melatonin
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample was taken to check for preoperative melatonin level. Plasma melatonin concentrations were measured using HPLC method in Inonu University Faculty of Pharmacy Analytical Chemistry Department research laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Endogenous Melatonin Levels — High Endogenous Melatonin Levels is Group 1 Low Endogenous Melatonin Levels is group 2

SUMMARY:
Interesting in living liver donor transplantation have greatly increased because of inadequacy of cadaveric organs and the inability to supply the growing need for cadaveric transplantation. Surgical procedures applied to living liver donors do not only physically demand organs, but can also cause psychological burden. It has been reported that melatonin had antioxidant, antinociceptive, hypnotic, anticonvulsant, neuroprotective, anxiolytic, sedative and analgesic properties. It was shown to administration of exogenous melatonin has been increase sedation and decrease anxiety in the preoperative period compared to placebo.

The aim of this study; To investigate preoperative and postoperative anxiety levels of CKV and to exam the relationship between anxiety levels and endogenous melatonin levels.

DETAILED DESCRIPTION:
Interesting in living liver donor (LLD) transplantation have greatly increased because of inadequacy of cadaveric organs and the inability to supply the growing need for cadaveric transplantation. Surgical procedures applied to LLD do not only physically demand organs, but can also cause psychological burden. Preoperative anxiety is seen in 60-80% of patients scheduled for surgery. It has been reported that melatonin had antioxidant, antinociceptive, hypnotic, anticonvulsant, neuroprotective, anxiolytic, sedative and analgesic properties. It was shown to administration of exogenous melatonin has been increase sedation and decrease anxiety in the preoperative period compared to placebo.

The aim of this study; To investigate preoperative and postoperative anxiety levels of LLD and to exam the relationship between anxiety levels and endogenous melatonin levels.

This prospective clinical study will perform at Inonu University Liver Transplant Institute. Anxiety of the patients included in the study will be measure with Spielberger State Anxiety Scale Scale (STAI FORM TX-1) in preoperative and postoperative period. It was designed to assess levels of state anxiety and traint anxiety, through 40 items scored by a likert-scale. Range of scores for each subtest is 20-80, the higher score indicating greater anxiety. A cut point of 39-40 has been suggested to detect clinically significant symptoms for the S-Anxiety scale. Patients without premedication will admit to the operating room. Before induction of anesthesia, the vascular access will perform and 3 mL of blood sample will take to check for preoperative melatonin level. Standard general anesthesia will perform to all donors. At the end of surgery, the patients will take to intensive care unit. After 24 hours, blood samples will take for post-melatonin. Plasma melatonin concentrations will measure using High Performance Liquid Chromatography (HPLC) method in Inonu University Faculty of Pharmacy Analytical Chemistry Department research laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Living liver donors, scheduled for right hepatectomy.
* between the ages of 18-65,
* American Society of Anesthesiologists Classification (ASA) 1-2

Exclusion Criteria:

* Patients with cardiovascular,
* neurological
* psychiatric disorders,
* opioid tolerance,
* sleep disturbance,
* hypnotic, neuroleptic, antidepressant, beta blocker and steroid use
* allergy history were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 Living liver donors (no= 60), between the ages of 18-65, ASA (American Society of Anesthesiologists Classification) 1-2 scheduled for right hepatectomy.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-02-15 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
The correlation between anxiety and melatonin levels | up to 24 hours
  Melatonin is a hormone secreted from the pineal gland. It shows a daily biorhythm. The circadian rhythm of melatonin changes according to age and it's production decreases with older ages. Melatonin level can be measured in the blood and in urine collected for 24 hours.It was designed to assess levels of state anxiety and traint anxiety, through 40 items scored by a likert-scale. the higher score indicating greater anxiety. A cut point of 39-40 has been suggested to detect clinically significant symptoms for the S-Anxiety scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu university, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altunkaya N, Erdogan MA, Ozgul U, Sanli M, Ucar M, Ozhan O, Sumer F, Erdogan S, Colak C, Durmus M. Changes in Melatonin, Cortisol, and Body Temperature, and the Relationship Between Endogenous Melatonin Levels and Analgesia Consumption in Patients Undergoing Bariatric Surgery. Obes Surg. 2018 Oct;28(10):3186-3192. doi: 10.1007/s11695-018-3313-x. PMID 29785473